CLINICAL TRIAL: NCT04849624
Title: Body Composition Study in Critically Ill Patients-Extended to COVID-19
Acronym: COVID-MUSCLE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: 2019615-7520-3
Record Dates: First submitted 2021-03-18; First posted 2021-04-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Covid19; Muscle Atrophy; Muscle Strength
MeSH Terms: conditions — Critical Illness; COVID-19; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICU COVID-19 patients: COVID-19 patients that are admitted into the ICU and fulfilled the eligibility criteria
  Interventions: Other: No Intervention
- ICU non-COVID-19 patients: Non-COVID-19 patients that are admitted into the ICU matched with ICU COVID-19 patients that are recruited and fulfilled the eligibility criteria
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study and involved no intervention

SUMMARY:
Muscle loss (ultrasound quadricep muscle) and muscle strength (handgrip and knee extension strength) will be compared between COVID-19 and non COVID-19 critically ill patients.

DETAILED DESCRIPTION:
Given the heightened inflammatory status among COVID-19 critically ill patients, we hypothesized that the rate of skeletal muscle loss is accelerated in this population, and this loss is even more pronounce than the general critically ill patients. We further hypothesized that the increased muscle loss will lead to worse functional outcome (lower muscle strength) in COVID-19 critically ill patients compared with age- and sex-matched non-COVID-19 critically ill patients, as it has been shown that quadriceps thickness is strongly correlated with functional status at ICU discharge. Furthermore, a recent systematic review and meta-analysis in survivors of coronavirus (severe acute respiratory syndrome, SARS or Middle-east respiratory syndrome, MERS, or COVID-19) also demonstrated reduced exercise capacity and quality of life at 6 months after hospitalization or ICU admission

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Admitted into the ICU due to COVID-19

Exclusion Criteria:

* Likely to transfer out from the ICU in 24 hours from screening
* Likely to die in the next 7 days
* Bedbound prior to hospital admission or bedbound in the hospital for >10 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 COVID-19 ICU patients as per the eligibility criteria will be recruited. A total of 20 non-COVID-19 ICU patients that are matched by age (+/- 10 years old), sex and ventilation mode (mostly will be with lung pathology) will be enrolled to compare their change in muscle mass and muscle strength at hospital discharge with COVID-19 ICU patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Rectus Femoris Thickness | Change in Rectus Femoris Thickness at day 7 or ICU discharge or hospital discharge compared with baseline (Day 1 of ICU admission)
  Change in Rectus Femoris Thickness
Rectus Femoris Cross-sectional Area | Change in Rectus Femoris Cross-sectional Area at day 7 or ICU discharge or hospital discharge compared with baseline (Day 1 of ICU admission)
  Change in Rectus Femoris Cross-sectional Area

SECONDARY OUTCOMES:
Forearm Muscle Thickness | Change in Forearm Muscle Thickness at day 7 or ICU discharge or hospital discharge compared with baseline (Day 1 of ICU admission)
  Change in Forearm Muscle Thickness
Handgrip Strength | Before Hospital Discharge
  BIlateral Handgrip Strength
Knee Extension Strength | Before Hospital Discharge
  BIlateral Knee Extension Strength

OTHER OUTCOMES:
Mortality | Mortality at day 28 (calculated from the first day of ICU admission)
  28-day Mortality
ICU length of stay | From date of enrolment until the date of discharged from the ICU, assessed up to 60 days
  Length of stay in the ICU
Hospital length of stay | From date of enrolment until the date of discharged from the hospital, assessed up to 60 days
  Length of stay in the Hospital
Length of Mechanical Ventilation | From date of commencement of mechanical ventilation until the date of liberation from mechanical ventilation, assessed up to 60 days
  Duration of Mechanical Ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee ZY, Ong SP, Ng CC, Yap CSL, Engkasan JP, Barakatun-Nisak MY, Heyland DK, Hasan MS. Association between ultrasound quadriceps muscle status with premorbid functional status and 60-day mortality in mechanically ventilated critically ill patient: A single-center prospective observational study. Clin Nutr. 2021 Mar;40(3):1338-1347. doi: 10.1016/j.clnu.2020.08.022. Epub 2020 Aug 28. PMID 32919818